CLINICAL TRIAL: NCT05318066
Title: Effect of a FLUid Bolus or a Low Dose VAsopressor Infusion on Cardiovascular Collapse Among Critically Ill Adults Undergoing Tracheal Intubation: a Randomized Controlled Trial (FLUVA Study)
Brief Title: Effect of a FLUid Bolus or a Low Dose VAsopressor Infusion on Cardiovascular Collapse Among Critically Ill Adults Undergoing Tracheal Intubation.
Acronym: FLUVA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3957; 3957 (Other: Tata Memorial Hospital)
Record Dates: First submitted 2022-03-22; First posted 2022-04-08 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Critically Ill Adults in the ICU, Requiring Endotracheal Intubation
MeSH Terms: interventions — Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: Randomization and treatment allocation All patients in ICU will be screened at the time the clinical team decides that tracheal intubation is required. Consent will be obtained from the patient's surrogate once they meet the inclusion and have no exclusion criteria. Once consent is obtained, the patient will be randomized.
  Study assignments will be placed in opaque randomization envelopes, and will be available to operators in the ICU. Study group assignment will remain concealed to study personnel and operators until after the decision has been made to enroll the patient in the study. The operator will open the next consecutively numbered envelope and follow the assignment of either fluid loading (FL arm) or low dose vasopressor (VP arm).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding Preparation for tracheal intubation will be done as per the ICU protocol * The airway operator will be blinded to the intervention and thus sent out of the patient's cubicle. The study team will administer a fluid bolus over 10 minutes. in the FL arm. No fluid will be administered in the VP arm. The fluid bag will be brought into the cubicle in a concealed bag. After fluid administration or not the fluid bag will be taken out in the same bag. A vasopressin infusion or saline infusion will be started at as per the assigned arm at the same time as the fluid bolus. The airway operator will enter the room and proceed with tracheal intubation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm Fluids (FL) (Active Comparator): 500 mL of ringer lactate over 10 minute prior to the administration of procedural medications.
  Interventions: Drug: Ringer Lactate and Norepinephrine infusion
- Arm Vasopressor (VP) (Active Comparator): Patients in this group would receive norepinephrine infusion at a dose of 0.08 μg/kg/min over 10 minutes prior and 5 minutes after tracheal intubation.
  Interventions: Drug: Ringer Lactate and Norepinephrine infusion

INTERVENTIONS:
Drug: Ringer Lactate and Norepinephrine infusion — Arm Fluids (FL)- 500 mL of ringer lactate over 10 minute prior to the administration of procedural medications.
  Arm Vasopressor (VP)- Patients in this group would receive norepinephrine infusion at a dose of 0.08 μg/kg/min over 10 minutes prior and 5 minutes after tracheal intubation.

SUMMARY:
Tracheal intubation, which is one of the most commonly performed procedures in the care of critically ill patients in intensive care unit, is associated with a high incidence of complications. Approximately 30% of emergent tracheal intubations in the ICU are associated with complications like hypotension, hypoxia, failed tracheal intubation, esophageal intubation, airway trauma, aspiration, cardiac arrest, and death. An observational study of tracheal intubation practices in critically ill patients across twenty-nine countries found cardiovascular instability to be the commonest among these adverse peri-tracheal intubation event.

Tracheal intubation performed in a controlled, non-emergent setting, is associated with few complications. However in ICU, conditions like underlying shock, respiratory failure, metabolic acidosis, and other patho-physiological changes contribute to the increased peri-tracheal intubation complications. Post tracheal intubation hypotension frequently occurs within a few minutes following tracheal intubation. The additive effects of hypovolemia, the suppression of the endogenous activation of sympathetic response by the anesthetics drugs as well as the intrathoracic positive pressure due to mechanical ventilation are implicated in this cardiovascular collapse after tracheal intubation in critically ill patients.

Post-tracheal intubation hypotension has been shown to be associated with higher in-hospital mortality and longer ICU and hospital length of stay. Hence patient optimization prior to tracheal intubation may be important to ensure hemodynamic stability to minimize further deterioration during tracheal intubation.

Few techniques to optimize hemodynamics before tracheal intubation commonly involve the use of intravenous fluids and vasopressor medications; however, there are no standards of care guiding these practices. Jaber et al included pre tracheal intubation fluid loading (isotonic saline 500 ml or starch 250 ml) as a part of tracheal intubation care bundle management to show improved outcomes. However it was an observational study and also it was not possible to evaluate the contribution of the individual hemodynamic components of the bundle given the concurrent implementation of other interventions.

And a recent study by Janz et al showed that pre loading with a 500-mL bolus of crystalloids before tracheal intubation did not identify any benefit. However this trial was stopped early for futility and moreover the volume of intravenous fluids that patients received before enrolment was not recorded.

Few trials have used vasopressor bolus prior to tracheal intubation to avoid post tracheal intubation hypotension or use of prophylactic use of vasopressors in preventing post spinal hypotension. However currently, there are no randomized trials or evidence-based guidelines to support the choice between fluid loading or vasopressors for the tracheal intubation of critically ill adults. We would like to conduct a randomised controlled study comparing the effects of fluid bolus or low dose vasopressor given prior to tracheal intubation on post tracheal intubation hypotension among critically ill adults.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary Objective:

Cardiovascular collapse - a composite endpoint defined as one or more of the following:

Decrease in systolic blood pressure (SBP) to less than 90 mm Hg or a decrease in mean arterial pressure to less than 65 mm Hg between induction and 5 min after tracheal intubation Cardiac arrest between induction and 1 hour after tracheal intubation; Death between induction and 1 hour after tracheal intubation

Secondary outcomes:

Clinical outcomes

* SBP <90 mm Hg or a MAP to less than 65 mm Hg within 5 min after tracheal intubation.
* Cardiac arrest between induction and 1 hour after tracheal intubation.
* Death between induction and 1 hour after tracheal intubation.
* Lowest SBP between induction and 5 min after tracheal intubation
* Ventilator-free days to 28 days
* ICU-free days to 28 days.
* Vasopressor free days at 28 days
* Need for Renal Replacement therapy post intubation in ICU
* ICU Mortality
* Hospital Mortality
* 28 Day Mortality

Safety outcomes

* Lowest arterial oxygen saturation between induction and 5 min after tracheal intubation.
* Incidence of hypoxaemia (oxygen saturation <90%) between induction and 5 min after tracheal intubation.
* Incidence of severe hypoxaemia (oxygen saturation <80%) between induction and 5 min after tracheal intubation.
* Incidence of hypertension (SBP >140) between induction and 5 min after tracheal intubation
* Oxygen saturation at 24 hours after tracheal intubation.
* Fraction of inspired oxygen at 24 hours after tracheal intubation.
* Pao2 /FiO2 ratio at 24 hours after tracheal intubation.

Process measures

* Initiation of an intravenous fluid bolus between induction and 5 min after tracheal intubation.
* Need for vasopressors in addition to study medication between induction and 5 min after tracheal intubation.
* Time from induction to successful tracheal intubation.
* Incidence of successful tracheal intubation on the first laryngoscopy attempt.
* Number of laryngoscopy attempts.
* Cormack-Lehane grade of glottic view on first attempt.
* Need for additional airway equipment or a second operator

Study design This is a pragmatic, single-centre, parallel group, randomised trial. comparing the impact of fluid loading vs low dose vasopressors on the incidence of cardiovascular collapse during tracheal intubation in critically ill adults.

STUDY SITES It will be conducted in 2ICUs (FICU and SICU) located at Tata Memorial Hospital, Mumbai.

Randomization and treatment allocation All patients in ICU will be screened at the time the clinical team decides that tracheal intubation is required. Consent will be obtained from the patient's surrogate once they meet the inclusion and have no exclusion criteria.Once consent is obtained, the patient will be randomized.

Study assignments will be placed in opaque randomization envelopes, and will be available to operators in the ICU. Study group assignment will remain concealed to study personnel and operators until after the decision has been made to enroll the patient in the study. The operator will open the next consecutively numbered envelope and follow the assignment of either fluid loading (FL arm) or low dose vasopressor (VP arm).

Blinding Preparation for tracheal intubation will be done as per the ICU protocol * The airway operator will be blinded to the intervention and thus sent out of the patient's cubicle. The study team will administer a fluid bolus over 10 minutes. in the FL arm. No fluid will be administered in the VP arm. The fluid bag will be brought into the cubicle in a concealed bag. After fluid administration or not the fluid bag will be taken out in the same bag. A vasopressin infusion or saline infusion will be started at as per the assigned arm at the same time as the fluid bolus. The airway operator will enter the room and proceed with tracheal intubation.

Study interventions Arm Fluids (FL)- 500 mL of ringer lactate over 10 minute prior to the administration of procedural medications.

Arm Vasopressor (VP)- Patients in this group would receive norepinephrine infusion at a dose of 0.08 μg/kg/min over 10 minutes prior and 5 minutes after tracheal intubation.

All medications that the patient is receiving for the critical illness will continue as usual during the study intervention period and be noted. Hypertension during study intervention period (defined as SBP greater than 140 mm Hg or more than 20 % of the baseline reading) will be managed by stopping the study drug infusion (norepinephrine or saline infusion). Treatment of hypertension will be left to the clinician's discretion. The study drug infusion will be resumed when blood pressure returns to its normal value up to 5 minutes after tracheal intubation. All study medications will continue for the patient as per the clinician's discretion. Hypotension during study intervention period (SBP, 90 mmHg or MAP <65) will be treated with a vasopressors or fluids as per the clinician's discretion.

Tracheal intubation Procedure Regardless of study group assignment, all airway operators will be encouraged to follow the institutional protocol for tracheal intubation. (Appendix 1) Monitors will be attached to the patient. Patient will be preoxygenation for 3 minutes, Rapid sequence tracheal intubation will be done using fentanyl, ketamine/ etomidate and rocuronium/Suxamethonium. Gentle bag mask is allowed if patient is at a risk for desaturation. Use of video laryngoscope and tracheal intubation aids will be encouraged. Tracheal intubation will be confirmed using capnography. Following confirmation of tube position and tube fixation the patient will be put on ventilator using protective lung ventilation.

Safety Intervention All complications that occur during the tracheal intubation procedure will be treated as per the clinician's discretion.

Data Collection:

All data collected are already a part of clinical data obtained in usual ICU care at the bedside or in the medical record. No additional data will be obtained beyond that which is obtained by bedside observation and from the electronic medical record. A trained, independent observer not involved in the performance of the procedure will collect data Demographic data

* Age
* Gender
* Height
* Weight
* BMI
* Acute Physiology and Chronic
* Health Evaluation (APACHE) II score
* Active medical problems at the time of tracheal intubation
* Active and chronic comorbidities complicating tracheal intubation
* Most recent pre-procedural Glasgow Coma Score
* Non-invasive ventilator and high flow nasal cannula use in the hour prior to starting pre-oxygenation.
* Pre intubation- PaO2, PCO2 and pH Tracheal intubation related data
* Indication for tracheal intubation
* Modality of pre-oxygenation
* Drugs used of induction with dose
* Drugs used for neuromuscular block with dose
* Use of ventilation between induction and laryngoscopy
* Laryngoscopy device used for first attempt
* Use of cricoid pressure,
* Cormack-Lehane grade of glottic view on the first attempt
* Use of a bougie or endotracheal tube with stylet on the first attempt
* Total number of attempts

Peri-procedural outcomes:

* Fluid volume received 4 hours prior to tracheal intubation
* Systolic blood pressure and oxygen saturation at the time of induction
* The lowest arterial oxygen saturation and systolic blood pressure from induction to 5 minutes after tracheal intubation
* The administration of a new fluid bolus between induction and 5 minutes after tracheal intubation
* The administration of a new dose of any vasopressor between induction and two minutes after tracheal intubation
* The total volume of new fluid bolus infused between induction and 5 minutes after tracheal intubation
* Post intubation PaO2, PCO2 and pH
* Any hypertension
* Any arrhythmia 0-1 hours:
* Cardiac arrest within 1 hour of tracheal intubation
* Death within 1 hour of tracheal intubation
* Systolic blood pressure, oxygen saturation, FiO2, and positive end expiratory pressure delivered every 5 minutes 1-24 hours:
* Systolic blood pressure, oxygen saturation, FiO2, and positive end expiratory pressure delivered every 1 hour

In-Hospital Outcomes:

* Total cumulative fluid administration in the ICU after randomization
* Date of extubation (ventilator-free days)
* Date of ICU discharge (ICU-free days)
* Date of death will be collected from the medical record.

STATISTICAL ANALYSIS Sample size estimation On the basis of previous research in our institute, the incidence of cardiovascular collapse in the fluid bolus group was found to be 40.5 %. Assuming this incidence rate and with the aim of reducing it by 50%, and to achieve a power of at least 80% with alpha error of 5% , 80 patients were needed in each group. Allowing for patients lost to follow up, 100 patients will be included in each group.

Analysis principles

* Primary analysis will be conducted on an intention-to-treat basis (patients with protocol violations are analyzed per the assigned treatment arm).
* All hypothesis tests will be two sided, with an α of 0.05 unless otherwise specified.
* All analyses will be unadjusted unless otherwise specified. SPSS Statistics (version 23.0) will be used for all analyses. Continuous variables will be reported as mean±SD or median and IQR; categorical variables will be reported as frequencies and proportions. All between-group comparisons with continuous variables will be performed using Mann-Whitney U tests and Fisher's exact test for categorical variables. Kaplan-Meier curves and log-rank tests will be used to analyze timeto-event comparisons between groups.

Primary analysis of the primary outcome The primary analysis will be an unadjusted, intention-to-treat comparison of patients randomised to the fluid bolus group versus patients randomised to the low dose vasopressor group with regard to the primary outcome of cardiovascular collapse. Between group differences will be tested using an unadjusted χ2 test. A p value <0.05 will be used to indicate statistical significance for the primary analysis.

Secondary analyses of the primary outcome To account for potential confounders, we will develop a logistic regression model with cardiovascular collapse (primary outcome) as the dependent variable and independent variables to include study group (fluid bolus group vs low dose vasopressors) and relevant confounders (age, Acute Physiology and Chronic Health Evaluation II (APACHE II) score at enrolment, presence of sepsis or septic shock and receipt of intravenous fluid infusion initiated prior to enrolment). We will also develop a logistic regression model accounting for the above variables plus any baseline characteristics that appear on visual review to be potentially imbalanced between the study groups.

Given the findings of the PrePARE trial subgroup analysis (ie, that the effect of fluid bolus administration on cardiovascular collapse may be related to the receipt of positive pressure ventilation during tracheal intubation), we will repeat the primary analysis excluding patients who did not receive positive pressure during l tracheal intubation.

Analysis of the secondary outcomes We will conduct unadjusted analyses examining the treatment effect of fluid loading on each of the pre-specified secondary and tertiary outcomes. Continuous outcomes will be compared with the Mann-Whitney U test and categorical variables with the Fischer exact test.

Handling of missing data Although we have allowed for loss to follow up in our power calculation, we do not anticipate that data for the primary outcome of cardiovascular collapse will be missing for any patients. Missing data will not be imputed for the primary or secondary outcome. In adjusted analyses, missing data for covariates may be imputed using a multiple imputation technique.

Ethics and dissemination Informed consent In current clinical practice, initiating an intravenous fluid bolus beginning prior to tracheal intubation and administering low dose vasopressors prior to tracheal intubation are both common management approaches, with significant variation between providers.15 . To be eligible for the trial, patients' treating clinicians must feel that initiation of a new fluid bolus for tracheal intubation is neither required nor contraindicated for the patient's optimal care. The protocol also states that vasopressor infusion will be stopped in case of hypertension. For these reasons, the trial is felt to pose minimal incremental risk compared with the clinical care patients would receive outside of the trial.

Tracheal intubation of critically ill adults is commonly an urgent or emergent procedure for which obtaining informed consent for the clinical procedure or informed consent for research is impracticable.

Information for patients and families A patient and family information sheet containing general study information and contact information for the research team provided to each patient and family at the time of admission to the study unit.

Adverse Events An adverse event is defined as any untoward medical occurrence in a clinical investigation where a participant is administered an intervention that does not necessarily have to have a causal relationship with the intervention. An adverse event therefore can be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an intervention, whether or not the incident is considered related to the intervention

A serious adverse event (SAE) is defined as any unexpected and untoward medical occurrence that is probably or possibly related to the study and meets any of the following criteria:

1. Results in death
2. Is life-threatening (defined as an event in which the participant was at risk of death at the time of the event and NOT an event that hypothetically might have caused death if it would have been more severe). Life-threatening cardiovascular complications, as defined as the primary endpoint of this trial, will be prospectively and systematically collected as the outcome. As such, these events will not be reported as SAEs. Similarly, life-threatening severe hypoxia will also be systematically collected as a secondary endpoint and will therefore not be reported as an SAE.
3. Requires inpatient hospitalization
4. Prolongs an existing hospitalization
5. Results in persistent or significant disability or incapacity
6. Results in a congenital anomaly or birth defect
7. Important medical event that requires an intervention to prevent any of a-f above.

   The Principal Investigator will be responsible for overseeing the safety of this trial on a daily basis. He will be available at any time for questions from the clinical team or bedside nurses, who will also be monitoring the patients continuously for adverse events and serious adverse events. Serious and unexpected adverse events potentially associated with study interventions will be recorded. As endotracheal tracheal tracheal intubation in the critical care setting is known to be independently associated with numerous adverse events including hypoxemia, aspiration, esophageal tracheal tracheal intubation, airway trauma, failed attempts at tracheal intubation, pneumothorax, pneumomediastinum, hypotension, severe bradycardia, cardiac arrest, and death, these events will be recorded as study outcomes and monitored to determine if a preponderance of adverse events in one study group merits consideration of stoppage of the trial. However, in the absence of an imbalance of the above events between study groups, these events are expected in the routine performance of the airway management procedure and will not be individually reported to the as serious and unexpected adverse events, unless the investigators or clinical team believe the event was related to the study intervention. As an additional safety measure, the exclusion criteria specifically state that airway management events in which urgency precludes performance of study or the operator foresees a potential need for or contraindication to manual ventilation between induction and tracheal intubation will not be included in the trial so all airway management events studied will be those in which the treating clinical team felt equipoise between the interventions being examined.

   Participant withdrawal and discontinuation criteria Withdrawal Criteria-
   1. Withdrawal of consent
   2. Following randomization, a clinician decides to limit therapy and hence not intubated the patient.

   Discontinuation Criteria

   1.Patient not tolerating the specific therapy. The reason and date of every withdrawal will be recorded in the patient study records. Follow up will be performed for all patients who discontinue due to an adverse event or any other safety parameter. Follow-up will also be performed for all patients who end participation in the protocol for another reason, but who also have an adverse event or other safety parameter that could have led to discontinuation. Follow-up will be conducted until the condition has resolved, until diagnosis of the adverse event or safety parameter is deemed chronic and stable, or as long as clinically appropriate. This follow-up will be documented in the patient study record as well.

   Privacy/Confidentiality Issues At no time during the course of this study, its analysis, or its publication will patient identities be revealed in any manner. The minimum necessary data containing patient or provider identities will be collected. All patients will be assigned a unique study ID number for tracking. Data collected from the medical record will be entered into the secure online database.

   Follow-up and Record Retention Patients will be followed after enrollment for 28 days or until hospital discharge, whichever occurs first. Data collected from the medical record will be entered into the secure online database. Hard copies of the data collection sheet completed at the time of the airway management event will be stored in a locked room until after the completion of enrollment and data cleaning. Once data are verified and the database is locked, all hard copies of data collection forms will be destroyed. All data will be maintained in the secure online database until the time of study publication.

   ANNEXURE 1 Criteria for endotracheal intubation

   These pre-determined criteria for endotracheal intubation and mechanical ventilation (MV) will be as follows to avoid delayed intubation:

   A) If participant shows at least any of the 2 following signs of persisting or worsening respiratory failure then he/she will be intubated
   1. a respiratory rate > 40 cycles/min
   2. lack of improvement of signs of respiratory-muscle fatigue
   3. development of copious tracheal secretions
   4. acidosis with a pH <7.25
   5. SpO2 < 90% for > 5min without technical dysfunction, or
   6. intolerance to NIV B) Or if participant shows any one of the following sign he/she will be intubated and receive mechanical ventilation

   <!-- -->

   1. hemodynamic instability defined by a SBP < 90 mmHg, MAP < 65 mmHg with requirement for vasopressor more than 0.25 mcg/kg/min
   2. deterioration of neurologic status with a Glasgow coma scale < 12 points

   ANNEXURE 2 PREPARATION OF TRACHEAL INTUBATION Preparation of equipment CO2-modul present and checked Patient equipped with pulse-oxymeter Box with regular intubation equipment present Box "difficult intubation" present Video laryngoscope Laryngoscope checked (light works) Reserve laryngoscope checked Bougie and stylet Magill forceps present Tube, cuff checked Reserve tube present Suction present and checked Facemask and bag present and checked Stethoscope present Material for tube-fixation present

   Preparation of drugs-The following drugs should be immediately available at bedside:

   Etomidate (2 mg/ml) Ketamine (2 mg/ml) Fentanyl (50 µg/ml) Midazolam (1 mg/ml) Succinylcholine (50 mg/ml) Rocuronium (10 mg/ml) Atropine (0.5 mg/ml) Ephedrine (5 mg/ml) Adrenaline (1 mg/ml and 0.1 mg/ml)

   ANNEXURE 3 RAPID SEQUENCE INTUBATION INSTITUTIONAL PROTOCOL After attaching monitors like ecg, pulse oximeter and non invasive bp monitor,one wide bore peripheral iv would be secured. Preoxygenation for at least 3mins will be performed in the high-risk patients with the help of NIV with an inspiratory pressure of 5-15 cm H2O, PEEP of 5 cm H2O and tidal volume of 6-8 mL/kg in a head-up position or with the help of HFNO. Apnoeic oxygenation will be considered to prolong safe apnoea time during intubation. After which total of 2 μg/kg intravenous fentanyl will be administered. Thereafter, an intravenous induction agent will be administered: etomidate 0.3 mg/kg or ketamine 2 mg/kg. The neuromuscular blocking drug Succinylcholine(1.5 mg/kg) or rocuronium (2 mg/kg) will be injected as soon as the injection of the induction agent is completed. Gentle bag mask is allowed if patient is at a risk for desaturation and is not full stomach. Use of cricoid pressure will be left upto the discretion of the clinician. Video laryngoscopy will be done after 45-60 sec after the injection of the neuromuscular blocking drug. Intubations will be performed using a rigid stylet loaded appropriate sized tracheal tube. Tracheal intubation will be confirmed by 6 continuous waveforms on capnography. Following confirmation of tube position and tube fixation the patient will be put on ventilator using protective lung ventilation

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old)
* Critically ill patients needing emergent tracheal intubation in ICU

Exclusion Criteria:

* Tracheal intubation performed in the out-of-ICU/hospital setting
* Tracheal intubation during cardiac arrest.
* Patients with age <18 years
* Elective tracheal intubation(for e.g for diagnostic/surgical procedures)
* Patients on vasoactive medications at the time of screening
* Hypotension (SBP <90) at screening
* Hypertension(SBP >140)at screening
* Urgency of tracheal intubation precludes performance of study procedures
* Operator feels administration of a fluid bolus vasopressor is strongly indicated or contraindicated
* Inability to obtain consent from the surrogate

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular collapse (composite outcome) | 1 hour
  Cardiovascular collapse - a composite endpoint defined as one or more of the following:
  Decrease in systolic blood pressure (SBP) to less than 90 mm Hg or a decrease in mean arterial pressure to less than 65 mm Hg between induction and 5 min after tracheal intubation. Cardiac arrest between induction and 1 hour after tracheal intubation. Death between induction and 1 hour after tracheal intubation.

SECONDARY OUTCOMES:
Hypotension | 28 days
  Systolic BP <90 mm Hg or a Mean Arterial Pressure to less than 65 mm Hg within 5 min after tracheal intubation.
Cardiac arrest | 1 hour
  Cardiac arrest between induction and 1 hour after tracheal intubation.
Death | 1 hour
  Death between induction and 1 hour after tracheal intubation.
Lowest Systolic Blood Pressure | 5 min
  Lowest SBP between induction and 5 min after tracheal intubation
Ventilator-free days to 28 days | 28 days
  Ventilator-free days to 28 days
ICU-free days to 28 days | 28 days
  ICU-free days to 28 days
Vasopressor free days at 28 days | 28 days
  Vasopressor free days at 28 days
Need for Renal Replacement therapy post intubation in ICU | 28 days
  Need for Renal Replacement therapy post intubation in ICU
ICU Mortality | No of days stayed in the ICU
  ICU Mortality
Hospital Mortality | No of days stayed in the Hospital
  Death during hospital stay
28 days Mortality | 28 days
  28 days Mortality
Lowest arterial oxygen saturation | 5 min
  Lowest arterial oxygen saturation between induction and 5 min after tracheal intubation.
Hypoxemia | 5 min
  Incidence of hypoxemia (oxygen saturation <90%) between induction and 5 min after tracheal intubation
Severe Hypoxemia | 5 min
  Incidence of severe hypoxemia (oxygen saturation <80%) between induction and 5 min after tracheal intubation
Incidence of hypertension | 5 min
  Incidence of hypertension (SBP >140) between induction and 5 min after tracheal intubation
Oxygen Saturation at 24 hours | 24 hours
  Oxygen saturation at 24 hours after tracheal intubation
FiO2 at 24 hours | 24 hours
  Fraction of inspired oxygen at 24 hours after tracheal intubation.
Pao2 /FiO2 ratio at 24 hours | 24 hours
  Pao2 /FiO2 ratio at 24 hours after tracheal intubation
Initiation of an intravenous fluid bolus | 5 min
  Initiation of an intravenous fluid bolus between induction and 5 min after tracheal intubation.
Need for vasopressors | 5 min
  Need for vasopressors in addition to study medication between induction and 5 min after tracheal intubation
Time from induction to successful tracheal intubation | 5 min
  Time from induction to successful tracheal intubation
Incidence of successful tracheal intubation on the first laryngoscopy attempt | 5 min
  Incidence of successful tracheal intubation on the first laryngoscopy attempt
Number of laryngoscopy attempts | 5 min
  Number of laryngoscopy attempts
Cormack-Lehane grade of glottic view on first attempt | 5 min
  Cormack-Lehane grade of glottic view on first attempt
Need for additional airway equipment or a second operator | 5 min
  Need for additional airway equipment or a second operator

CONTACTS AND LOCATIONS:
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India